CLINICAL TRIAL: NCT05481970
Title: Opioid Free Anesthesia for Upper Limb Surgery in Obese Patients.
Brief Title: Opioid Free Anesthesia in Obese Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Rana Ahmed Abdelghaffar, Lecturer of anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: opioid free anesthesia
Record Dates: First submitted 2022-07-20; First posted 2022-08-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2022-07

CONDITIONS: Opioid Free Anesthesia
Keywords: opioid free anesthesia; obese; dexmedetomidine; ketamine
MeSH Terms: conditions — Obesity | interventions — Dexmedetomidine; Dexamethasone; Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Active Comparator): Group A , Induction of general anesthesia will be done using lidocaine (1.5 mg/kg), propofol (2-3 mg/kg), and atracurium (0.5 mg/kg). Dexmedetomidine 0.5 µg/kg over 10 min, started 10 min before induction. Following tracheal intubation, dexmedetomidine infusion generally will be initiated at 0.6 μg/kg/h and titrated between 0.2 and 1.0 μg/kg/h according to the heart rate maintaining bispectral index (BIS) between 40-60, lidocaine (1.5 mg/kg/h). ketamine will be given as a bolus dose of 0.3 mg/kg after induction and prior to skin incision then 0.2 mg/kg/h as an infusion. Patients will receive dexamethasone (8 mg i.v.) after induction.
  Interventions: Drug: dexmedetomidine,ketamine,lidocaine,propofol
- Opioid group (Placebo Comparator): In group (B) (OBA) for induction of anesthesia, patients will receive propofol 2-3mg/kg, fentanyl 1-2mcg/kg and atracurium 0.5 mg/kg as a muscle relaxant to facilitate intubation. Fentanyl bolus doses of 0.5-1 mcg/kg will be given to keep BIS score 40-60 during surgery.
  Interventions: Drug: fentanyl,propofol

INTERVENTIONS:
Drug: dexmedetomidine,ketamine,lidocaine,propofol — Group (A): Induction of general anesthesia will be done using lidocaine (1.5 mg/kg), propofol (2-3 mg/kg), and atracurium (0.5 mg/kg). Dexmedetomidine 0.5 µg/kg over 10 min, started 10 min before induction. Following tracheal intubation, dexmedetomidine infusion generally will be initiated at 0.6 μg/kg/h and titrated between 0.2 and 1.0 μg/kg/h according to the heart rate maintaining bispectral index (BIS) between 40-60, lidocaine (1.5 mg/kg/h). ketamine will be given as a bolus dose of 0.3 mg/kg after induction and prior to skin incision then 0.2 mg/kg/h as an infusion. Patients will receive dexamethasone (8 mg i.v.) after induction.
  Other Names: dexamethasone
  Arms: Dexmedetomidine group
Drug: fentanyl,propofol — In group (B) for induction of anesthesia, patients will receive propofol 2-3mg/kg, fentanyl 1-2mcg/kg and atracurium 0.5 mg/kg as a muscle relaxant to facilitate intubation. Fentanyl bolus doses of 0.5-1 mcg/kg will be given to keep BIS score 40-60 during surgery.
  Other Names: fentanyl
  Arms: Opioid group

SUMMARY:
Using opioids in the clinical practice of anesthesia was astonishing. They are good analgesics and used widely to modulate perioperative pain, but analgesia with these drugs can be associated with many side effects that may lead to prolongation of hospital stay and recovery period like respiratory depression, delirium, impaired gastrointestinal function, urine retention, post-operative nausea and vomiting (PONV), and addiction. The most significant opioid side effect is respiratory depression. This is especially important in patients suffering from obesity. Obese patients already have a restrictive lung disease leading to decrease in functional residual capacity and total lung compliance. Anesthetics and analgesics specially opioids make these respiratory problems become worse with increasing the incidence of hypoxia. These side effects can be avoided by using opioid free anesthesia (OFA) techniques.

Opioid free anesthesia recently become more applicable and popular in different centers, it provides pain control with marked reduction in opioid consumption. However, researches and studies still unable to explore definite explanations or techniques regarding it. The base of OFA is that not only one drug can replace opioids. It is a multimodal anesthesia. Multiple drugs are used to achieve it. They are hypnotics,N-methyl-D-aspartate (NMDA) antagonists (ketamine, magnesium sulfate), sodium channel blockers (local anesthetics), anti-inflammatory drugs (NSAID, dexamethasone), and alpha-2 agonists (dexmedetomidine, clonidine). Regional anesthesia and nerve blocks also have a role. In this study, using OFA the investigators are hoping to achieve a good quality of care to obese patients helping in fast track surgery with less complications and so shorter period of hospital stay

DETAILED DESCRIPTION:
Patients will be randomly allocated (by closed envelope method) to two groups:

Group A (n=38) will have opioid free anesthesia (OFA) Group B (n=38) will have opioid based anesthesia (OPA) All patients will be subjected to a preoperative clinical examination and routine preoperative laboratory investigations. Patients also will be trained on how to deal with the VAS score before surgery. The visual analog scale (VAS) is a pain score using a 10-cm line with two ends "no pain" on the left end and the "worst pain" on the right end, used to track pain for a patient or to compare pain between patients.(9,10) In the operating room (OR), peripheral oxygen saturation (spo2), noninvasive blood pressure and electrocardiogram ( ECG) will be monitored and recorded as a baseline reading. A peripheral intravenous cannula will be inserted t hen patients in both groups will receive 1mg of midazolam prior induction of anesthesia. Preoxygenation 3-5 minutes before induction will be done. Group (A): Induction of general anesthesia will be done using lidocaine (1.5 mg/kg), propofol (2-3 mg/kg), and atracurium (0.5 mg/kg). Dexmedetomidine 0.5 µg/kg over 10 min, started 10 min before induction. Following tracheal intubation, dexmedetomidine infusion generally will be initiated at 0.6 μg/kg/h and titrated between 0.2 and 1.0 μg/kg/h according to the heart rate maintaining bispectral index (BIS) between 40-60, lidocaine (1.5 mg/kg/h). ketamine will be given as a bolus dose of 0.3 mg/kg after induction and prior to skin incision then 0.2 mg/kg/h as an infusion. Patients will receive dexamethasone (8 mg i.v.) after induction. In group (B) for induction of anesthesia, patients will receive propofol 2-3mg/kg, fentanyl 1-2mcg/kg and atracurium 0.5 mg/kg as a muscle relaxant to facilitate intubation. Fentanyl bolus doses of 0.5-1 mcg/kg will be given to keep BIS score 40-60 during surgery.

All Patients will be mechanically ventilated with 50% O2 and 50% air and the end-tidal carbon dioxide( CO2) will be maintained between 30 - 35 mmHg. Anesthesia will be maintained by isoflurane and atracurium 0.1-0.2 mg/kg every 20-30 minutes. Reversal of muscle relaxants will done by using intravenous neostigmine (0.05 mg/kg) and atropine (0.01 mg/kg) at the end of surgery and the patient will be extubated when the patient will be able to breath spontaneously with tidal volume ≥5ml/kg and spo2>92%. Paracetamol 1gm i.v. infusion and ketorolac 30 mg slow i.v injection will be used at the end of surgery and before emergence in both groups. At the recovery room, patients will assess their pain and rating it using VAS score, monitored for postoperative pain, the patients will leave the post anesthesia care unit (PACU) with Aldrete score more than 9. (11) Any patient with Vas score ≥4, will receive tramadol 1mg/kg i.v. with a maximum dose 600mg/day.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status Ⅱ , Ⅲ.
* body mass index (BMI) ≥30 kg/m2.
* Have upper limb surgeries (orthopedics, plastic,…) under general anesthesia.

Exclusion Criteria:

* Known allergy to the drugs will be used in the study.
* Pregnancy and lactation.
* Addiction or recent use of opioids'
* Patients will not be able deal with visual analog score(VAS).
* Hepatic, Renal and cardiac diseases in advanced stages.
* History of epilepsy or seizures.
* Patients with cerebrovascular disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Attacks of postoperative pain with vas score ≥4 | 24 hours postoperative
  The visual analog scale (VAS) is a pain score using a 10-cm line with two ends "no pain" on the left end and the "worst pain" on the right end, postoperative pain with vas score ≥4 will be monitored and recorded
rescue doses of tramadol | 24 hours postoperative
  time of rescue doses of tramadol
how many rescue doses of tramadol | 24 hours postoperative
  number of rescue doses of tramadol

SECONDARY OUTCOMES:
Hypoxia | every 2hours for 24 hours.
  number of patients with hypoxia (an Spo2 level of less than 95%)
Postoperative nausea and vomiting. | 24 hours postoperative
  Postoperative nausea and vomiting( number of attacks)
Postoperative usage of antiemetics | 24 hours postoperative
  number of patients who will need rescue dose of antiemetic medication.
Intraoperative bradycardia | intraoperative
  number of patients who will develop intra-operative bradycardia HR≤50bpm,
Intraoperative hypotension | intraoperative
  number of patients who will develop intra-operative hypotension mean arterial blood pressure ( mABP) ≤60 millimetre of mercury (mmHg)
Intraoperative hypertension | intraoperative
  number of patients who will develop intra-operative hypertension mABP ≥90mmHg).
ICU admission. | 24 hours postoperative
  number of participants who will need intensive care unit
extubation time | 60 minutes after cessation of anesthesia
  time when endotracheal tube removed from the patients

CONTACTS AND LOCATIONS:
Overall Officials: Rana A Abelghaffar, MD, Principal Investigator — Faculty of medicine , Fayoum university
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No